CLINICAL TRIAL: NCT00262743
Title: A Phase I/II Study of Daily Oral Polyphenon E in Asymptomatic, Rai Stage 0-II Patients With Chronic Lymphocytic Leukemia
Brief Title: Green Tea Extract in Treating Patients With Stage 0, Stage I, or Stage II Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454773; P30CA015083 (NIH); 1155-05 (Other: Mayo Clinic IRB); NCI-2009-01227 (Registry Identifier: NCI-CTRP); MC0419 (Other: Mayo Clinic Cancer Center); NCT00166335 (obsolete NCT alias)
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Leukemia
Keywords: B-cell chronic lymphocytic leukemia; stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — polyphenon E

ARMS (1):
- polyphenon E (Experimental): Designed to assess toxicity, treatment response, and pertinent laboratory measurements in patients with previously untreated, asymptomatic, Rai Stage 0-II CLL.
  Interventions: Biological: Polyphenon E

INTERVENTIONS:
Biological: Polyphenon E — Phase I Dose Escalation:. 400 mg orally twice a day to 2000 mg orally twice a day
  Phase II: 2000 mg orally twice a day

SUMMARY:
RATIONALE: Green tea extract contains ingredients that may slow the growth of certain cancers.

PURPOSE: This phase I/II trial is studying the side effects and best dose of green tea extract and to see how well it works in treating patients with stage 0, stage I, or stage II chronic lymphocytic leukemia (CLL).

DETAILED DESCRIPTION:
OBJECTIVES:

Phase I

* Determine the maximally tolerated dose of green tea extract (Polyphenon E) in patients with previously untreated stage 0-II chronic lymphocytic leukemia.
* Describe the dose-limiting toxicity of green tea extract (Polyphenon E).

Phase II

* Evaluate the response rate and response duration of patients with previously untreated, asymptomatic Rai stage 0-II chronic lymphocytic leukemia treated with green tea extract (Polyphenon E) for 6 months at the MTD.
* Further characterize toxicity.

OUTLINE: This is a phase I, dose-escalation study of green tea extract (Polyphenon E) followed by a phase II study.

* Phase I: Patients receive oral green tea extract (Polyphenon E) once or twice daily for 4 weeks. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of green tea extract (Polyphenon E) until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive green tea extract (Polyphenon E) as in the phase I portion of the study at the MTD.

After completion of study treatment, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 73 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of chronic lymphocytic leukemia (CLL)

  * Stage 0, I, or II disease
  * Previously untreated disease
  * Splenomegaly, hepatomegaly, or lymphadenopathy are not required for the diagnosis of CLL
  * Absolute lymphocyte count > 10,000/mm^3
  * Lymphocytosis must consist of small to moderate size lymphocytes, with ≤ 55% prolymphocytes, atypical lymphocytes, or lymphoblasts morphologically
  * Phenotypically characterized B-CLL defined by all of the following criteria:

    * A population of leukemic cells that co-expresses the B-cell antigen CD23 as well as CD5 in the absence of other T-cell markers (CD3, CD2, etc.)
    * Dim surface immunoglobulin expression
    * Exclusively κ or λ light chains
  * Mantle cell lymphoma must be excluded by demonstrating the absence of the t(11:14) by FISH testing
* Patients who require chemotherapy for treatment of CLL, based on any of the following criteria, are excluded:

  * CLL-related symptoms requiring treatment, including any of the following:

    * Unintentional weight loss ≥ 10% body weight within the previous 6 months
    * Extreme fatigue
    * Fevers > 100.5°F for 2 weeks without evidence of infection
    * Night sweats without evidence of infection
  * Evidence of progressive marrow failure due to CLL involvement of bone marrow as manifested by the development of worsening anemia (hemoglobin < 11 g/dl) and/or thrombocytopenia (platelet count < 100,000/mm^3)

    * Thrombocytopenia due to immune phenomena (ITP) is permitted as long as platelet count is ≥ 100,000/mm^3and the patient is not on active pharmacologic therapy
  * Massive (i.e. > 6 cm below left costal margin) or progressive splenomegaly
  * Massive nodes or clusters (i.e., > 10 cm in longest diameter) or progressive adenopathy
  * Progressive lymphocytosis with an increase of > 50% over 2 month period, or an anticipated lymphocyte doubling time of < 6 months

PATIENT CHARACTERISTICS:

* Platelet count ≥ 100,000/µL
* ANC ≥ 1500/µL
* Hemoglobin ≥ 11 g/dL
* Total or direct bilirubin ≤ 1.5 x upper limit of normal (ULN)
* AST (SGOT) and ALT (SGPT) ≤ 2 x ULN
* Creatinine ≤ 1.5 x ULN OR creatinine clearance ≥ 40 mL/min
* May have a history of autoimmune hemolytic anemia (AIHA) and positive Coombs test provided there has not been active hemolysis requiring transfusion or steroid treatment ≤ 10 weeks prior to registration
* ECOG performance status 0, 1, or 2
* Life expectancy of ≥ 6 months
* No uncontrolled infection
* No myocardial infarction within the past 6 weeks
* No New York Heart Association class III or IV congestive heart failure
* Not pregnant or nursing
* Negative pregnancy test
* Must employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], or abstinence, etc.) prior to study entry and for the duration of study participation
* No other severe medical or psychiatric illness
* No active hemolysis requiring transfusion or other pharmacologic therapy

PRIOR CONCURRENT THERAPY:

* At least 8 weeks since prior and no other concurrent over the counter green tea or green tea extract
* No prior daily use of over the counter green tea products for medicinal purposes for > 4 weeks (phase II only)
* No other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-FDA-approved indication and in the context of a research investigation)
* No concurrent combination anti-retroviral therapy for HIV positive patients
* No concurrent oral steroid preparations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2005-08; Primary Completion 2010-05 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tait D. Shanafelt, MD, Study Chair — Mayo Clinic; Jose F Leis, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Result] Shanafelt TD, Call TG, Zent CS, LaPlant B, Bowen DA, Roos M, Secreto CR, Ghosh AK, Kabat BF, Lee MJ, Yang CS, Jelinek DF, Erlichman C, Kay NE. Phase I trial of daily oral Polyphenon E in patients with asymptomatic Rai stage 0 to II chronic lymphocytic leukemia. J Clin Oncol. 2009 Aug 10;27(23):3808-14. doi: 10.1200/JCO.2008.21.1284. Epub 2009 May 26. PMID 19470922
- [Result] Shanafelt TD, Call TG, Zent CS, Leis JF, LaPlant B, Bowen DA, Roos M, Laumann K, Ghosh AK, Lesnick C, Lee MJ, Yang CS, Jelinek DF, Erlichman C, Kay NE. Phase 2 trial of daily, oral Polyphenon E in patients with asymptomatic, Rai stage 0 to II chronic lymphocytic leukemia. Cancer. 2013 Jan 15;119(2):363-70. doi: 10.1002/cncr.27719. Epub 2012 Jul 3. PMID 22760587

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 73 participants were enrolled at the Mayo Clinic from August 2005 - October 2009.
Pre-assignment Details: Thirty-six (36) and 37 patients recruited to the phase I and phase II portions, respectively. Three phase I patients were replaced and one patient was ineligible for evaluation. Per study design, the 36 eligible phase II participants along with the 6 phase I participants treated at the phase II dose level were evaluated (n=42).
Groups:
- Phase I Polyphenon E: Dose ranging from 400 to 1,800 mg orally twice a day for 6 months
- Phase II Polyphenon E: 2000mg orally twice daily for 6 months
Period: Overall Study
Arm/Group | Phase I Polyphenon E | Phase II Polyphenon E
Started | 27 | 42
Completed | 27 | 30
Not Completed | 0 | 12
Not completed — Adverse Event | 0 | 9
Not completed — Disease progression | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Phase I Polyphenon E: Dose ranging from 400 to 1,800 mg orally twice daily for 6 months
- Phase II Polyphenon E: 2000mg twice daily for 6 months
- Total: Total of all reporting groups
Arm/Group | Phase I Polyphenon E | Phase II Polyphenon E | Total
Number analyzed (Participants) | 27 | 42 | 69
Age Continuous [Median (Full Range); unit: years] | 62 [44 to 76] | 60 [41 to 78] | 60 [41 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 18 | 30 | 48
Region of Enrollment [Number; unit: participants]
  United States | 27 | 42 | 69
Dose Level of Polyphenon E [Number; unit: participants]
  400 mg | 3 | 0 | 3
  800 mg | 6 | 0 | 6
  1000 mg | 3 | 0 | 3
  1200 mg | 6 | 0 | 6
  1400 mg | 3 | 0 | 3
  1600 mg | 3 | 0 | 3
  1800 mg | 3 | 0 | 3
  2000 mg | 0 | 42 | 42
Fluorescence In Situ Hybridization (FISH) Abnormalities [Number; unit: participants] — This test determines the presence of abnormalities in specific chromosomes of CLL cells, which are associated with more or less aggressive forms of cancer. Patients with abnormalities of chromosome 11 (deletion 11q23) and 17 (deletion 17p13) experience rapid progression of their CLL.
  participants
    Normal | 6 | 10 | 16
    deletion (13q14.2) | 17 | 27 | 44
    Trisomy 12 | 4 | 4 | 8
    deletion (11q23) | 0 | 1 | 1
Rai Stage [Number; unit: participants] — Rai staging is a way to categorize the disease progression of chronic lymphocytic leukemia (CLL); higher stages reflect increasing severity.
  Rai Stage 0: Lymphocytosis only, Rai Stage I: Lymphocytosis and lymphadenopathy, Rai Stage II: Lymphocytosis and hepatomegaly +/- splenomegaly
  participants
    Stage 0 | 15 | 13 | 28
    Stage I | 8 | 24 | 32
    Stage II | 4 | 5 | 9
ZAP-70 Status [Number; unit: participants] — This test is used to predict the rate of progression from diagnosis to need for treatment in CLL. Participants with positive ZAP-70 (>=20%) tend to experience a more aggressive course of CLL.
  participants
    Positive (>=20%) | 6 | 12 | 18
    Negative (<20%) | 21 | 30 | 51
CD38 Status [Number; unit: participants] — This test is used to predict the rate of progression from diagnosis to need for treatment in CLL. Participants with positive CD38 (>=30%) tend to experience a more aggressive course of CLL.
  participants
    Positive (>=30%) | 4 | 7 | 11
    Negative (<30%) | 23 | 35 | 58
Immunoglobulin Variable Heavy Chain (IGVH) Mutation Status [Number; unit: participants] — IGVH testing helps predict which patients will experience a more aggressive (if the gene is unmutated, <=2%) or less aggressive (if the gene is mutated, >2%) course of CLL. This technically complex test is only available at select medical institutions.
  participants
    Unmutated (<=2%) | 7 | 6 | 13
    Mutated (>2%) | 18 | 27 | 45
    Unavailable | 2 | 9 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Confirmed Response [Complete Response (CR) and Partial Response (PR)] on 2 Consecutive Evaluations at Least 4 Weeks Apart
Description: National Cancer Institute working group criteria (NCIWG) was used to assess response.
  * CR: no lymphadenopathy, hepatomegaly, splenomegaly or constitutional symptoms; normal complete blood count; confirmed by bone marrow (BM) aspirate & biopsy
  * PR: 50% decrease in peripheral blood lymphocytes, lymphadenopathy, liver/spleen size, presence/absence of constitutional symptoms; plus ≥1 of the following: ≥1500/μL polymorphonuclear leukocytes, >100000/μL platelets, >11.0 g/dL hemoglobin or 50% improvement for these parameters without transfusions
Time Frame: 6 months
Population: Phase II participants who satisfied all eligibility criteria, signed the consent form and started therapy were evaluated for this endpoint.
Measure: Number; unit: participants
Arm/Group | Phase II Polyphenon E
Number analyzed (Participants) | 42
participants | 1

2. Primary Outcome: Number of Participants With Biological Response (Bio-R) on 2 Consecutive Evaluations at Least 4 Weeks Apart
Description: Bio-R: A reduction in the absolute lymphocyte count (ALC) of more than 20% from the pretreatment level for at least 2 months or a >= 30% reduction in all palpable lymphadenopathy without meeting the NCIWG criteria for PR was required
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Phase II Polyphenon E
Number analyzed (Participants) | 42
participants | 28

3. Secondary Outcome: Number of Participants With a Confirmed Complete Response (CR)
Description: A confirmed complete response is a CR which is reported on 2 consecutive cycles at least 4 weeks apart. CR is defined in Primary Outcome Measure #1.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Phase II Polyphenon E
Number analyzed (Participants) | 42
participants | 0

4. Other Pre Specified Outcome: 24 Month Treatment Free Survival Rate
Description: Percentage of participants who were alive and treatment (for progressive CLL) free at 24 months. The 24 month treatment free survival, with 95% CI, was estimated using the Kaplan-Meier method.
Time Frame: 24 months (from registration)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II Polyphenon E
Number analyzed (Participants) | 42
percentage of participants | 79 [62 to 92]

ADVERSE EVENTS:
Arm/Group | Phase II Polyphenon E
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 40/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II Polyphenon E (N=42)
Hemoglobin decreased (Blood and lymphatic system disorders) | 12 (27)
Vision blurred (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 12 (21)
Abdominal pain (Gastrointestinal disorders) | 20 (37)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 29 (68)
Dyspepsia (Gastrointestinal disorders) | 12 (24)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 15 (32)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 27 (71)
Vomiting (Gastrointestinal disorders) | 5 (5)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 22 (59)
Fever (General disorders) | 1 (1)
Flu-like symptoms (General disorders) | 10 (12)
Hypersensitivity (Immune system disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Alanine aminotransferase increased (Investigations) | 22 (57)
Alkaline phosphatase increased (Investigations) | 6 (30)
Aspartate aminotransferase increased (Investigations) | 19 (32)
Blood bilirubin increased (Investigations) | 4 (13)
Creatinine increased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 5 (11)
Platelet count decreased (Investigations) | 15 (34)
Anorexia (Metabolism and nutrition disorders) | 14 (25)
Blood glucose increased (Metabolism and nutrition disorders) | 7 (18)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 3 (8)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (5)
Dizziness (Nervous system disorders) | 5 (6)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 13 (21)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (6)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes